CLINICAL TRIAL: NCT05533645
Title: Development and Validation of a Food Frequency Questionnaire to Assess Sodium Intake in Hospitalized Patients or in Medical Consultation
Brief Title: Food Frequency Questionnaire to Assess Sodium Intake
Acronym: EVALSEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021_0523; 2022-A00241-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Renal Insufficiency
Keywords: natriuresis; Hypertension; Renal insufficiency; Sodium; Table salt
MeSH Terms: conditions — Hypertension; Renal Insufficiency | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): patients with high blood pressure or chronic kidney diseases stages 4-5
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — These patients complete the food frequency questionnaire in order to validate it for lower sodium consumptions. The experimental group has already received dietary advices regarding salt consumption during during their recent consultations.

SUMMARY:
EvalSel can precisely assess the salt intake of hospitalized patients in nephrology and cardiology or in medical consultation. It can determine salt consumption to the nearest gram.

The objectives of this food frequency questionnaire are to arrive at a precise dietary diagnosis and to quickly identify the dietary errors made by the patients.

EvalSel is useful for doctors to quickly obtain an assessment of the salt consumption of their patients, so they can refer them to dietitians if necessary. It can be used on the day of admission to hospital or during medical follow-ups to know the evolution of their consumption over the long term and improve their care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high blood pressure, CKD stages 4-5 and patients free from any diseases
* Patients over 18 years old
* Patients in nephrology and cardiology consultation or recruited by CIC
* Patients with health insurance
* Patients willing to follow the full study

Exclusion Criteria:

* Loss of salt by vomiting, diarrhea or sweating (intense sport or intense fever 3 days before urine collection) which can cause a decreasing natriuresis
* Modification of the therapeutic management of patients during the study period
* Taking certain drugs like effervescent drugs, Gaviscon and Tolvaptan during the day of urine collection, as well as diuretics (unless they are taken long-term and the diuresis is stable) which can cause an increasing natriuresis
* Pregnant or breastfeeding women
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intra-class correlation coefficient between the quantitative measurement of sodium consumption and the 24-hour natriuresis measurement and verification of the 24-hour creatininuria values | through study completion an average of 18 months
  Intra-class correlation coefficient between the quantitative measurement of sodium consumption by the EvalSel questionnaire and the 24-hour natriuresis measurement (amount of sodium in 24-hour urine) and verification of the 24-hour creatininuria values (amount of creatinine in 24-hour urine) to confirm that the urine collection was performed correctly.

CONTACTS AND LOCATIONS:
Overall Officials: d GUYONNET, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Huriez - Service Endocrinologie Diabétologie, Lille, France